CLINICAL TRIAL: NCT05619510
Title: Testing an Intervention to Reduce Pain and Depression Among Older Women With Physical Disabilities
Brief Title: Pain Reduction Through Empowered Recovery (PRIME) Study
Acronym: PRIME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00341962; P30AG022845 (NIH)
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Pain, Chronic; Depressive Symptoms; Depression; Disability Physical
MeSH Terms: conditions — Chronic Pain; Depression

STUDY DESIGN:
Intervention Model Description: A wait list control group will be used for this study. Participants will be randomized to either the intervention group or the wait list control group. Participants in the intervention group will start the intervention immediately. Participants in the wait list control will start after 2-3 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The data collectors, interventionists, and investigator will be masked to which group participants belong to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait List Control Group (Other): This group will be randomized to wait list control. They will serve as a control for the intervention at time points 1 and 2. However after a 2-3 month period they will receive the intervention.
  Interventions: Behavioral: PRIME Intervention
- Intervention Group (Experimental): Individuals randomized to this group will start the intervention immediately and have outcomes measured at three time points.
  Interventions: Behavioral: PRIME Intervention

INTERVENTIONS:
Behavioral: PRIME Intervention — Participants who are randomized to the intervention will participate in five virtual or in person visits with a nurse where the nurse uses self regulation theory as a guide to help them set their own goals surrounding pain and depression and use tailored strategies to address these goals. The second component will include six virtual Acceptance Commitment Therapy (ACT) sessions, led by a clinical psychologist. There will be 3-5 other research participants in the sessions.

SUMMARY:
Chronic pain and depression or low mood are often experience by women who age with or into disabilities. Due to various factors women with disabilities often experience this cycle of pain and depression. Both of these conditions can be debilitating and lead to declines in health. Treating these conditions simultaneously, particularly , in older adults can be complicated due to side effects, risks of poor access to pain management and mental health care , and complications from other co occuring conditions. In order to address this cycle in older women with disabilities the investigators are testing the Women in Pain Reduction through Improved Mood and Empowerment (PRIME) study. The PRIME intervention includes four in person visits by a nurse to the women's homes where the participants set goals regarding pain and depression and the nurse helps the participants strategize ways to meet these goals. The second component of the study will be eight group sessions virtually with other participants in the study. The group sessions will be led by a clinical psychologist who will engage in Acceptance Commitment Therapy with the women.

DETAILED DESCRIPTION:
Chronic pain and depression frequently co-occur among older women with disabilities, and each can exacerbate the other in a worsening cycle. This co-occurrence may be due, in part, to pain and depression sharing biologic etiologies such as inflammation. Beyond each individual category of risk, the intersection of age, sex, and disability place older women with disabilities at even higher risk of having co-occurring pain and depression.There are several effective multi-component behavioral interventions for either pain or depression, but not both outcomes in combination, and none were designed to integrate social determinants of health to address the inequities inherent in being an older woman with disabilities. Addressing these two conditions in this population warrants multicomponent interventions that are appropriate for and inclusive of all older women with disabilities. The proposed study is to apply self-regulation theory to refine and further test the feasibility of a tailored behavioral activation intervention, older women with disabilities in Pain Reduction through Improved Mood and Empowerment (PRIME) Study Aim 1: Leveraging the investigators previous research, the investigators will enroll 15-30 community dwelling women , ages 50 and over, with physical disabilities , living in Maryland who have pain and depression in the Women in PRIME clinical trial.

Aim 2: The investigators will determine a) feasibility and acceptability of the intervention and b) if strategies and evaluation techniques are appropriate.

ELIGIBILITY:
Inclusion Criteria:

* self-reported pain >4 out of a 0-10 scale that has lasted longer than 3 months and prohibits at least one valued or daily activity,
* physical disability based on the 2008 American Community Survey. The survey includes one question about disability in the following categories: sensory, physical, self-care, ability to go outside of the home, and independent living difficulty. Candidates who report having mobility disabilities will be considered for the study,
* non-institutionalized and living in Maryland, and
* score a 5 or higher on the PHQ9 (depression measure) at least two times during a two week period (screening call and then at first data collection visit via video)
* 50 years of age and older, 6) female

Exclusion Criteria:

* hospitalized > 3 times in the last year,
* participating in physical therapy,
* have a terminal diagnosis (<1 year expected survival),
* > moderate intellectual impairment (5-7 errors) based on the Short Portable Mental Status Questionnaire (SPMSQ), 81 and
* unable to understand or speak English. We will exclude anyone with more than three hospitalizations and/or have a terminal diagnosis because of the acuity of their conditions which may limit the effectiveness of the intervention. Physical therapy may impact the outcomes of the intervention and having impaired cognition may make it difficult for participants to engage in the nurse visits, set goals and participate in the ACT sessions.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-03-16 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain intensity measure | Baseline, 12 weeks, 24 weeks
  Pain Intensity will be measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain intensity measure. PROMIS Pain Intensity is a 3 question measure with a range of 3-15 with a higher score indicating increased pain intensity.
Change in Pain Interference as assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline, 12 weeks, 24 weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS) pain interference is a 6 question measure with a range of 6-30 with a higher score indicating increased pain interference.
Change in Pain Behavior as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS)Pain behavior measure | Baseline, 12 weeks, 24 weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS) pain interference is a 20 question measure with a range of 20-100 with a higher score indicating increased pain behaviors
Change in Depression as assessed by the Patient Health Questionnaire 9 (PHQ9) | Baseline, 12 weeks, 24 weeks
  The Patient Health Questionnaire 9 (PHQ9) measures depressive symptoms. The score range is 0-27 with a higher score indicating more severe depression.
Change in depression as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) 57 | Baseline, 12 weeks, 24 weeks
  The Patient Reported Outcomes Measurement System (PROMIS)57 the Patient Reported Outcomes Measurement Information System (PROMIS) 57, which is includes an 8-item instrument that can be used to measure self-reported negative mood, view of self, and somatic symptoms. The score range for PROMIS 57 is 8-40. Higher scores indicate more depressive symptoms

SECONDARY OUTCOMES:
Change in Psychological Flexibility as assessed by the Psychological Flexibility in Pain Instrument | Baseline, 12 weeks, 24 weeks
  The Psychological Flexibility in Pain Instrument will be used. The ability to act in alignment of goals, values and in acceptance while living with pain and distress.The Psychological Inflexibility in Pain Scale (PIPS) is a 12-item scale measuring avoidance of pain, and fusion with pain thoughts. Scores range from 7-84 with a higher score indicating increased psychological inflexibility in pain.
Change in Interleukin-6 (IL-6), Interleukin-8 (IL-8), and | Baseline and 12 weeks
  All three IL-6, IL-8, tumor necrosis factor (TNF) and will be on a cytokine panel that will be measured using sweat patches. The unit of measurement used will be picograms per millimeter (pg/ml) .
Change in Goal Attainment as assessed by self report | At baseline and at 12 weeks
  Self-report if goals were achieved fully, partially or not at all
Change in Comorbidities as assessed by the Charlson Comorbidity Index (CCI) | Baseline and 12 weeks
  The Charlson Comorbidity Index will be used to obtain a score for number of chronic conditions from 19 categories.The CCI consists of 19 selected conditions that are weighted and summed to an index on a 0-33 scale. Higher scores indicate more comorbidities.
Change in Sleep Disturbance as assessed by the 4 item PROMIS sleep disturbance measure | Baseline and 12 weeks
  Sleep disturbance will be measured using the 4 item PROMIS sleep disturbance measure. This six item scale is used to measure sleep disturbances in the past 7 days and the range is 6 -30 with higher scores indicating more sleep disturbances.
Communication with Health Care Providers- Patient Reaction Assessment | Baseline and 12 weeks
  The Patients' Reaction Assessment has a 5-item subscale used to measure perceived ability to communicate with providers. The sub scale on perceived ability to communicate with providers can have scores ranging from 0-35 with higher scores indicating higher perceived ability to communicate.

CONTACTS AND LOCATIONS:
Overall Officials: Janiece L Taylor, PhD, Principal Investigator — Johns Hopkins School of Nursing; Elaine Wethington, PhD, Study Chair — Cornell Roybal Center (Weill Cornell Medicine)
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

REFERENCES:
- [Result] Taylor JL, Drazich BF, Roberts L, Okoye S, Rivers E, Wenzel J, Wright R, Beach MC, Szanton SL. Pain in low-income older women with disabilities: a qualitative descriptive study. J Women Aging. 2020 Jul-Aug;32(4):402-423. doi: 10.1080/08952841.2020.1763895. Epub 2020 May 31. PMID 32475259
- [Result] Drazich BF, Jenkins E, Nkimbeng M, Abshire Saylor M, Szanton SL, Wright R, Beach MC, Taylor JL. Exploring the Experiences of Co-morbid Pain and Depression in Older African American Women and Their Preferred Management Strategies. Front Pain Res (Lausanne). 2022 Feb 28;3:845513. doi: 10.3389/fpain.2022.845513. eCollection 2022. PMID 35295801
- [Derived] Taylor JL, Clair CA, Atkins S, Wang C, Booth A, Reid MC, Wethington E, Regier NG. A protocol for a wait list control trial of an intervention to improve pain and depressive symptoms among middle-aged and older women living with disabilities. Contemp Clin Trials. 2025 Mar;150:107826. doi: 10.1016/j.cct.2025.107826. Epub 2025 Jan 28. PMID 39884648

DOCUMENTS (1):
  • Informed Consent Form (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT05619510/ICF_000.pdf